CLINICAL TRIAL: NCT00367289
Title: CT for Diagnosis of Implant Stability in Revision Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Leonid Kandel, Hadassah Medical Organization
Other Study IDs: ctosteolysis-HMO-CTIL
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2006-08

CONDITIONS: Hip Arthroplasty; Knee Arthroplasty; Osteolysis
MeSH Terms: conditions — Osteolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
All patients over 18 who undergo a revision of hip or knee arthroplasty will be included. Patients undergo a CT of the hip joint. A radiologist will mark the presence of cysts and bone loss and will assess implant stability.

After the surgery, the surgeon will fill a similar form.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for hip or knee revision arthroplasty
* age over 18

Exclusion Criteria:

* fractures
* dislocations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Revision hip and knee arthroplasty patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Kandel, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel